CLINICAL TRIAL: NCT06634641
Title: Assessment of Clozapine-related Immunodeficiency Effect in Parkinsons Disease Patients
Brief Title: Clozapine-related Immunodeficiency in Parkinsons Disease
Acronym: CLOZIDPD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2024_843_0069
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Clozapine; Parkinson's Disease (PD); Immunodeficiency; Psychosis
Keywords: clozapine; parkinson's disease; immunodeficiency; psychosis
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Psychotic Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood test — Only carrying out additional immunological assays during blood tests before initiation of treatment, six months after initiation of treatment and then one year after initiation of treatment.

SUMMARY:
Clozapine is a second generation antipsychotic drug used in psychiatry to treat schizophrenia, affective disorders or certain symptoms of dementia. In neurology, clozapine is frequently used and recommended to manage symptoms of psychosis associated with Parkinson's disease (PD). The risk of neutropenia or agranulocytosis associated with clozapine estimated at 1.3% is well known to doctors around the world with a peak at one month and a decrease in risk after more than a year of treatment. This risk has led to the policy of "no blood, no drugs" and monitoring of the complete blood count (CBC) weekly for 18 weeks and then monthly for the duration of treatment.

Some studies suggest an increased risk of infections related to immunodeficiency induced by clozapine itself. This clozapine-induced immunodeficiency would be comparable to that encountered in patients with common variable immunodeficiency or under immunosuppressive treatment. In addition, this immunosuppressive effect linked to clozapine would not be dose dependent but time dependent. However, the only studies currently performed have been in psychiatric patients treated for schizophrenia.

It seems important to specifically explore clozapine-related immunodeficiency in PD patients treated with clozapine for PD-related psychosis. In this study, the investigators propose to evaluate the variations in serum immunoglobulin levels and lymphocyte subpopulations (B, T, NK) in parkinsonian patients treated with Clozapine at 6 months and 1 year after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old with Parkinson's disease according to MDS 2015 criteria
* Psychotic symptoms requiring treatment with Clozapine
* Patients with initially a normal leukocyte count (number of white blood cells

  ≥ 3500/mm3 [3.5 x 109/l] and an absolute neutrophil count PNN ≥ 2000/mm3 [2 x 109/l])
* patients in whom the number of white blood cells (WBC) and the absolute number of neutrophils (PNN) may be determined regularly at the following intervals: once a week during the first 18 weeks of treatment and, thereafter, at least every 4 weeks for the duration of the treatment. This monitoring must be continued throughout the treatment and for 4 weeks who follow the complete cessation of CLOZAPINE
* Informed and written consent.
* Affiliation to a social security system

Exclusion Criteria:

* Patients with a contraindication to the use of Clozapine according to the summary of product characteristics (SPC)
* Hypersensitivity to the active substance or to any of the excipients.
* Patients who cannot receive regular blood tests.
* History of granulopenia or toxic or idiosyncratic agranulocytosis (unless it results from previous chemotherapy).
* History of agranulocytosis induced by CLOZAPINE
* Treatment with CLOZAPINE should not be started at the same time as substances known to have a high potential for inducing agranulocytosis; The concomitant administration of depot antipsychotics is not recommended.
* Functional bone marrow failure.
* Uncontrolled epilepsy.
* Alcoholic or induced psychosis, drug intoxication, comatose states.
* Circulatory collapse and / or CNS depression regardless of the aetiology.
* Severe renal or cardiac disorders (eg: myocarditis).
* Active liver disease with nausea, anorexia or jaundice; progressive liver disease, liver failure.
* Paralytic ileus.
* Patient with another potential cause of immunosuppression
* Immunosuppressive or immune modulatory treatment active or stopped for less than 5 years
* Anti-epileptic treatment active or stopped for less than 5 years
* Chemotherapy active or stopped for less than 5 years
* Solid or hematologic cancer active or treated for less than 5 years
* Human immunodeficiency virus infection
* Already known constitutional immune deficiency
* Nephrotic syndrome
* Protein-losing enteropathy
* A history of radiotherapy
* Long-term use of corticosteroids
* Patient with potentially major cognitive disorders defined by a MoCA score less than or equal to 23
* Pregnant or breastfeeding women
* Patient under guardianship/curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
change in serum IgG levels | 6 months
  change in serum IgG levels after 6 months of clozapine treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Salouël, France

IPD SHARING:
Plan to Share IPD: No